CLINICAL TRIAL: NCT00675987
Title: Protocol Merck 318-00: A Double-Blind, Placebo-Controlled, Randomized, Parallel, Clinical Trial To Study The Effect Of Losartan Potassium On Endothelial Dysfunction And Insulin Resistance In Obese Patients With Impaired Fasting Glucose
Brief Title: A Randomized Clinical Trial To Study Losartan On Endothelial Dysfunction and Insulin Resistance In Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Mark Alan Creager, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2007-P-000490
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Hypertension; Hyperglycemia
Keywords: Impaired Fasting Glucose FPG >100-<126 mg/dL
MeSH Terms: conditions — Obesity; Hypertension; Hyperglycemia | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Losartan (Active Comparator): Losartan 100 mg 1 tab po QD
  Interventions: Drug: losartan
- Placebo (Placebo Comparator): Placebo 1 tab po QD
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: losartan — losartan 100 mg tablets 1 tab po QD
  Other Names: Cozaar
  Arms: Losartan
Drug: Placebo control — Placebo 1 po QD
  Arms: Placebo

SUMMARY:
The main purposes of this study are to find out if the study drug losartan (Cozaar) or placebo ("sugar pill") has an effect on insulin sensitivity (how your body responds to insulin) and to measure the effect of the study drug losartan or placebo on how the arteries in your arm dilate (enlarge to carry more blood).

We hope to learn if taking losartan changes the amount of certain proteins in the blood that effect blood vessel function.

Losartan is approved by the US FDA to treat high blood pressure. It will take approximately 4 months for you to complete this study.

ELIGIBILITY:
Inclusion Criteria:

* Currently taking 1 or no antihypertensive medication
* Male and female between 18 and 75 years of age
* Mean trough sitting diastolic blood pressure (SiDBP) ≥80 and < 100 mm Hg
* Mean trough sitting systolic blood pressure (SiSBP) ≥120 and <160 mm Hg
* Non-diabetic patients with fasting plasma glucose ≥100 mg/dL and <126 mg/dL
* Body mass index (BMI) >30 and <40
* Waist circumference >40 inches in males, > 35 inches in females
* A patient who is of reproductive potential and agrees to remain abstinent or use acceptable methods of birth control (intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, condom, hormonal contraception, vasectomy) within the projected duration of the study

Exclusion Criteria:

* Secondary hypertension of any etiology (renal artery stenosis, coarctation of the aorta or pheochromocytoma, hypertension induced by oral contraceptives)
* History of malignant hypertension
* Any clinically significant renal disease including single functioning kidney, and known history of anuria. Any severe renal impairment, as manifested by serum creatinine more than 1.5 mg/dL, or proteinuria >2+ by urine dipstick
* Known sensitivity or intolerance to angiotensin II receptor antagonists
* Type I or II diabetes
* Inability or unwillingness to abstain from taking prohibited medications during the study period
* History of myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG), congestive heart failure (CHF), unstable angina, transient ischemic attack (TIA), or cerebrovascular accident (CVA)
* Concomitant cardiac conditions that would make it unsafe to participate in the trial (e.g., clinically significant atrioventricular (AV) conduction disturbance, atrial flutter, atrial fibrillation, potentially life-threatening ventricular arrhythmias, decompensated valvular disease, presence of hemodynamically significant obstructive valvular disease, or cardiomyopathy)
* History of angioedema and/or organ damage from hypertension
* Serum potassium < 3.5 or > 5.5 mEq/L
* Any clinically significant laboratory value which in the investigator's judgment could be clinically significant to the outcome of this study.
* History of clinically important gastrointestinal resection or malabsorption
* Patient with a history or current evident of any condition, therapy, lab abnormality, or other circumstance that might confound the results of the study, or interfere with the patient's participation for the full duration of the study, such that it is not in the best interest of the patient to participate. (Including but not limited to: recent or current alcoholism, drug abuse within the prior 2 years, mental or legal incapacitation, any disease which could reasonably be expected to be fatal or life-threatening, or a history of malignancy ≤ 5 years prior to signing informed consent.)
* Currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent.
* Inability to be taken off all current antihypertensive medication and placed on placebo for up to 12 weeks.
* Unwillingness or unlikely to adhere to the study procedures, keep appointments, or is planning to relocate during the study.
* Arm circumference great than 52 cm
* Smokers or former smokers who have quite less than 1 year prior to Visit 1
* Anemia (Hemoglobin < 11)
* Allergy to latex
* Deformed hands and/or fingers that would interfere with the collection of pulse volume amplitude measurements
* History of Raynaud's disease or any other vascular condition
* Bilateral mastectomy
* Aortic stenosis
* Patient is taking high doses of antioxidant supplements (vitamins, minerals, or other)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Creager, MD, Principal Investigator — Brigham and Women's Hospital
Locations (9):
- United States (9):
  - CAVS Clinical Research Center, Little Rock, Arkansas
  - VA San Diego Health Care System, San Diego, California
  - University of Miami Diabetes Research Institute, Miami, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Brigham and Women's Hospital Cardiovascular Division, Boston, Massachusetts
  - St. Lukes Roosevelt Hospital, New York, New York
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - University of Texas SW Medical Center at Dallas, Dallas, Texas
  - Hypertension Clinical Pharmacology Baylor Clinic, Houston, Texas

REFERENCES:
- [Result] Perlstein TS, Henry RR, Mather KJ, Rickels MR, Abate NI, Grundy SM, Mai Y, Albu JB, Marks JB, Pool JL, Creager MA. Effect of angiotensin receptor blockade on insulin sensitivity and endothelial function in abdominally obese hypertensive patients with impaired fasting glucose. Clin Sci (Lond). 2012 Feb;122(4):193-202. doi: 10.1042/CS20110284. PMID 21861845

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan 100 mg 1 Tab po QD: Losartan 100 mg 1 tab po QD
- Placebo 1 Tab po QD: Placebo 1 tab po QD
Period: Overall Study
Arm/Group | Losartan 100 mg 1 Tab po QD | Placebo 1 Tab po QD
Started | 26 | 27
Completed | 26 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan 100 mg 1 Tab po QD | Placebo 1 Tab po QD | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 27 | 53
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (10.5) | 53.8 (8.3) | 52.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 12 | 15 | 27
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity Utilizing the Euglycemic Hyperinsulinemic Clamp
Description: Insulin clamp derived insulin sensitivity, as insulin stimulated glucose disposal corrected for steady state insulin level.
Time Frame: baseline, 8 weeks
Population: analysis was ITT, but limited to those with interpretable data (3 clamp studies were excluded)
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 27 | 26
mg/kg/min | 5.3 (4.5) | 2.8 (1.7)

2. Primary Outcome: Insulin Sensitivity Utilizing Endothelial Function as Assessed by Pulse Volume Amplitude
Description: Endothelial function assessed as the ratio of pulse volume amplitude after compared with before a reactive hyperemia stimulus, measured by peripheral (fingertip) arterial tonometry. Reported values indicate the percentage change from Baseline in the ratio of pulse volume amplitude after compared to before the reactive hyperemia stimulus.
Time Frame: baseline, 8 weeks
Population: analysis was ITT, but limited to those with interpretable data (3 clamp studies were excluded)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 27 | 26
percentage change | 1.76 (0.7) | 2.11 (0.7)

3. Secondary Outcome: Change in Urine Albumin/Creatine
Description: Urine was obtained to assess for the presence of microalbuminuria.
Time Frame: baseline, 8 weeks
Population: 27 participants were randomized to placebo, and 26 participants were randomized to Losartan, but 1 placebo participant and 1 Losartan participant did not complete the study.
Measure: Mean (95% Confidence Interval); unit: mg/mmol
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 26 | 25
mg/mmol | 0.4 [-0.1 to 0.9] | 0.2 [-0.3 to 0.8]

4. Secondary Outcome: Change in hsCRP (High-sensitivity C-reactive Protein)
Description: hsCRP (high-sensitivity C-reactive protein) is a marker of inflammation
Time Frame: baseline, 8 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 26 | 25
percentage change | -10 [-32 to 20] | -34 [-50 to -13]

5. Secondary Outcome: Change in VCAM-1(Vascular Cell-adhesion Molecule-1)
Description: VCAM-1 is an immunoglobulin-like adhesion molecule expressed on activated endothelial cells.
Time Frame: baseline, 8 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 26 | 25
ng/ml | 29 [-20 to 79] | -21 [-70 to 28]

6. Secondary Outcome: Change in MCP-1 (Monocyte Chemoattractant Protein-1)
Description: MCP-1 is one of the key chemokines that regulate migration and infiltration of monocytes/macrophages.
Time Frame: baseline, 8 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 26 | 25
pg/ml | -37 [-80 to 6.8] | -24 [-65 to 18]

7. Secondary Outcome: Change in Ox-LDL (Oxidized Low-density Lipoprotein)
Description: ox-LDL measures protein damage due to the oxidative modification of the ApoB subunit on LDL cholesterol.
Time Frame: baseline, 8 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units/l
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 26 | 25
units/l | -2.0 [-8.1 to 4.1] | -5.5 [-11.9 to 0.9]

8. Secondary Outcome: Change in F2-isoprostanes
Description: F2-isoprostanes is a marker of oxidative stress.
Time Frame: baseline, 8 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: ng/mg of creatinine
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 26 | 25
ng/mg of creatinine | 0.4 [-0.9 to 1.6] | 0.9 [-0.4 to 2.2]

9. Secondary Outcome: Change in E-selectin
Description: E-selectin is expressed on inflamed endothelial cells in response to treatment with inflammatory cytokines.
Time Frame: baseline, 8 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 26 | 25
ng/ml | -1.6 [-4.5 to 1.3] | -0.6 [-3.5 to 2.3]

ADVERSE EVENTS:
Arm/Group | Losartan | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No